CLINICAL TRIAL: NCT05353010
Title: Open-Label, 1-Sequence, 2-Period, Multiple Oral Dose Phase 1 Study to Evaluate Effect of IN-A001 on Pharmacokinetics of Tacrolimus in Healthy Volunteers
Brief Title: A Study to Evaluate Effect of IN-A001 on Pharmacokinetics of Tacrolimus in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IN_APA_120
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Period 1: A; Period 2: B and C (Experimental): A: Oral Administration of Tacrolimus 5mg once / B: Oral Administration of IN-A001(Tegoprazan) 50mg QD for 7 days / C: Oral Administration of IN-A001(Tegoprazan) 50mg + Tacrolimus 5mg once
  Interventions: Drug: Tacrolimus; Drug: IN-A001(Tegoprazan); Drug: IN-A001(Tegoprazan) + Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus 5mg (1 mg * 5 capsules)
  Other Names: prograf
Drug: IN-A001(Tegoprazan) — IN-A001 50mg(Tegoprazan 50mg* 1 tablet)
  Other Names: K-CAB
Drug: IN-A001(Tegoprazan) + Tacrolimus — IN-A001 50mg(Tegoprazan 50mg*1 tablet) and Tacrolimus 5mg(1mg * 5capsules)
  Other Names: IN-A001: K-CAB, Tacrolimus: Prograf

SUMMARY:
This study aims to investigate the effect of IN-A001 50mg on the pharmacokinetics of Tacrolimus 5mg in healthy volunteers

DETAILED DESCRIPTION:
This is a open-label, 1-sequence, 2-period, multiple oral dose, phase 1 study. Healthy subjects will be assigned to a group and sequentially administerd Tacrolimus and IN-A001.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index(BMI) ≥ 19.0 and ≤ 28.0 kg/m^2 at the time of screening.
2. Those who agreed to use combination of effective or medically approved contraceptive method from the date of first administration of investigational product(IP) to the end of the clinical trial (when testing for final safety evaluation).
3. In the case of female participant, who has negative result at the hCG urine pregnancy test and is not pregnant or currently breastfeeding.

Exclusion Criteria:

1. Has clinically significant infections
2. Has a history of malignancy
3. Has a history of gastrointestinal disease that may affect the absorption of investigational product.
4. Has genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose absorption disorder etc.
5. History of hypersensitivity and severe allergic reaction to any of the components of IP.
6. Has participated in any other clinical study, etc. and received IPs within 180 days prior to the screening visit.
7. Excessive smoking (> 10 cigarettes/day) within 14 days prior to the screening visit.
8. Excessive drinking ((> 21 units/week) within 14 days prior to the screening visit.
9. Has shown the following results from the laboratory test during the screening period.

   * AST, ALT level > 1.5 × ULN at screening;
   * eGFR(estimated glomerular filtration rate) estimated on the basis of CKD-EPI is less than 60 mL/min/1.73 m2;
10. Has shown the following results during the 12-lead electrocardiogram during the screening period.

    * QTc > 450 ms
    * Clinically significant abnormal rhythm and findings when the investigator medically determines
11. Determined ineligible for study participation by the investigator for other reasons.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Cmax of Tacrolimus | up to 72 hours(period 1), up to 240 hours(period 2)
  Maximum Plasma Concentration at Steady State of Tacrolimus
Tmax of Tacrolimus | up to 72 hours(period 1), up to 240 hours(period 2)
  Time to Cmax at steady state
AUClast of Tacrolimus | up to 72 hours(period 1), up to 240 hours(period 2)
  Area under the concentration-time curve from dosing (time 0) to the time of the last measured concentration
AUCinf of Tacrolimus | up to 72 hours(period 1), up to 240 hours(period 2)
  Area under the curve from time 0 extrapolated to infinite time
T1/2β of Tacrolimus | up to 72 hours(period 1), up to 240 hours(period 2)
  Half-life of the drug during elimination phase

SECONDARY OUTCOMES:
Point estimates and 90% CI for log (GMR of Period 2 Cmax, AUClast, AUCinf) / log (GMR of Period 1 Cmax, AUClast, AUCinf) of Tacrolimus | up to 72 hours(period 1), up to 240 hours(period 2)
  log(GMR of Period 2 Cmax, AUClast, AUCinf) / log (GMR of Period 1 Cmax, AUClast, AUCinf)
Cmax of Tegoprazan | up to 240 hours(period 2)
  Maximum Plasma Concentration at Steady State of Tegoprazan
Tmax of Tegoprazan | up to 240 hours(period 2)
  Time to Cmax at steady state
AUClast of Tegoprazan | up to 240 hours(period 2)
  Area under the concentration-time curve from dosing (time 0) to the time of the last measured concentration
AUCinf of Tegoprazan | up to 240 hours(period 2)
  Area under the curve from time 0 extrapolated to infinite time
T1/2β of Tegoprazan | up to 240 hours(period 2)
  Half-life of the drug during elimination phase

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea